CLINICAL TRIAL: NCT02913859
Title: Hormone Therapy With or Without Definitive Radiotherapy in Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Ana Frobe, MD, PhD, Prof., University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHSestre
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; hormone-sensitive; metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic radiotherapy (Experimental): long-term hormonal therapy (LHRH agonist and/or antiandrogens) plus radiotherapy to the pelvis and prostate
  Interventions: Radiation: Radiotherapy to the pelvis; Drug: Hormonal therapy (LHRH agonist and/or antiandrogens)
- No pelvic radiotherapy (Active Comparator): long-term hormonal therapy ( LHRH agonist and/or antiandrogens) alone
  Interventions: Drug: Hormonal therapy (LHRH agonist and/or antiandrogens)

INTERVENTIONS:
Radiation: Radiotherapy to the pelvis — Radiotherapy to the pelvis and prostate
  Arms: pelvic radiotherapy
Drug: Hormonal therapy (LHRH agonist and/or antiandrogens) — life-long hormonal therapy (LHRH agonist and/or antiandrogens)
  Other Names: medical castration and/or antiandrogens

SUMMARY:
PART I

Hormone therapy with or without definitive radiotherapy in metastatic prostate cancer

The goal of this clinical study PART I is to determine impact of radiotherapy treatment in combination with standard androgen deprivation therapy comparing with androgen deprivation therapy alone at controlling metastatic prostate cancer. The primary objective: to determine disease progression free survival in man with metastatic (M1) prostate cancer (PC) undergoing androgen deprivation therapy with or without definitive radiotherapy of the primary tumor.The secondary objective: to determine disease progression (local, bone marrow, visceral) in men with metastatic prostate cancer (M1PC) undergoing systemic therapy with/without definitive radiotherapy of the primary tumor, to determine expression in number of genes analysed 8: 2 housekeeping genes; integrin subunits αv, β3, β5, α4β1 ; 3 EMT markers N-cadherin, E-cadherin, vimentin before radiotherapy, after radiotherapy and at the time of the disease progression , to determine plasma serotonin (5HT, 5 hydroxytryptamine). Subgroup analysis in locally advanced prostate cancer (serves as a control group for integrins analysis): to determine expression in number of genes analysed 8: 2 housekeeping genes; integrin subunits αv, β3, β5, α4β1 ; 3 epithelial-mesenchymal transition (EMT) markers N-cadherin, E-cadherin, vimentin before radiotherapy, after radiotherapy and at the time of the disease progression.

PART II

Identification of genetic determinants of disease progression and castrate resistance in metastatic prostate cancer.

The goal of this clinical study PART II is to assess feasibility of genomic testing in the multidisciplinary clinical management of metastatic prostate cancer, to gain insight in specific genomic signature(s) of progressive metastatic prostate cancer in the natural course of disease spanning from primary tumor to metastases, to test if 'treatment selection' and/or 'treatment adaptation' as means of evolutionary pressures represent the mechanistic models of castrate resistance and ultimate treatment failure following course of androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
PART I

Standard therapy for men presenting with metastatic prostate cancer is initiation of androgen suppression, whereas radiotherapy or surgery are currently used only in palliative efforts to relieve symptoms of bleeding, pain, or obstruction. The integration of radiation to the prostate has not been prospectively explored in the metastatic setting.

Although there is no study evidence on the effect of local therapy on outcomes in metastatic prostate cancer, there are hypotheses-generating data that support this concept as an appropriate question to be answered in the context of a randomized trial. Prospective data show improved outcomes for men with locally advanced prostate cancer undergoing multimodality therapy with androgen-deprivation therapy (ADT) or radiation therapy (RT) compared to systemic monotherapy alone . Continuing on the spectrum of the disease, recent data presented at the 2014 European Society for Medical Oncology Annual Meeting showed improved failure-free survival in men with clinically positive lymph nodes receiving combination ADT and RT versus ADT alone.

Several population-based studies have shown improved overall survival in men with metastatic disease undergoing combination local and systemic therapy versus standard-of-care systemic therapy alone .

Previous studies showed that initial event at a metastatic site is not the arrival of tumor cells but rather the clustering of bone marrow-derived cells . This cells make the local microenvironment of the secondary organ more receptive to tumor cell colonization and are stimulated by endocrine factors released by the primary tumor . According to this, local treatment of the primary tumor could postpone the formation and the growth of distant metastases; metastatic prostate cancer may represent a heterogeneous population and the impact of local treatment on disease progression on survival might be influenced by primary tumor characteristics.

Many studies support the importance of integrins in prostate cancer development and progression by promoting proliferation, invasion and metastasis. Targeting specific integrins and their matrix interaction may provide a way to prevent metastatic bone prostate cancer.

Serotonin or 5-hydroxytryptamine (5-HT) is a well-known neurotransmitter that mediates a wide variety of physiological effects. An increase in the number of 5-HT-releasing neuroendocrine (NE) cells has been correlated with prostate tumor progression. However, it is particularly unclear whether released 5-HT or the release of 5-HT has a role in tumor cell growth .

Serotonin is a well-known mitogen which mediates a wide variety of physiological effects via multiple receptors, of which receptor subtype 1 (5-HTR1) has been identified in prostate cancer (PC) cell lines. Recently, 5-HT has been found to show growth-promoting activity and to be functionally related to oncogenes .

Previous studies showed that 5-HT stimulated the proliferation of prostate cancer cells mediated by 5-HT receptors 5-HTR1A and R1B and the secretion system of prostate NE cells is capable of 5-HT synthesis and metabolism plays a significant role in prostate tumor generation and progression. These findings are crucial for the development of potential drugs to slow prostate tumor progression.

PART II

Genomic alternations leading to development of metastasis, treatment resistance and ultimate disease progression include multistep mutational events on androgen signalling axis, in tumor suppressor genes and oncogenes and finally DNA repair defects which are currently being intensively studied using large multinational collaborative efforts (Robinson Cell 2015, PCF Stand up to Cancer West Coast Dream Team). Despite this growing body of data on biology behind the different phenotypes of metastatic prostate cancer seen in clinic, little is known on how discovery of specific gene/pathway involved in multi-step process of disease progression impact clinical decisions, especially in limited resource setting. Furthermore, there is a knowledge gap addressing the impact of ADT, which is mainstay of the treatment of metastatic prostate cancer, on mutational landscape in the context of hormone sensitive disease. For programs starting to embrace personalised treatment paradigm it is essential to gain insight how to integrate genomic data in the clinic and even more, to test whether genomic testing in the course of disease of patient with metastatic prostate cancer is feasible.

Primary goal of this PART II study is to assess feasibility of genomic testing in the pilot group of five patients with prostate cancer who develop metastases from the large pool of patients with prostate cancer followed prospectively in our multidisciplinary clinic. Secondary goal is to determine level of genomic instability and principal mutational events in the metastases as opposed to the primary tumor, with addition of differentiating genomic outlook of metastases before and after emergence of castrate resistant disease.

(i) Aims 1, 2, 3: To assess feasibility of genomic testing in the critical steps in management of the patient with metastatic prostate cancer and to characterise genomic signature of progressive metastatic prostate cancer

In prospectively followed cohort of participants with prostate cancer, participants who develop metastatic disease will be identified, and approached for genomic testing before initiation of ADT. The investigators plan to characterize the genomics of metastatic prostate cancer using whole exome sequencing for single nucleotide variations (SNVs), gene rearrangements (GRs) and copy number variants/alternations (CNVs). Eligible participants are those who develop measurable and biopsiable metastatic disease (i.e. lymph nodes or bone lesion) that is detected using classical radiological staging methods (bone scan, computerized tomography) regardless of underwent primary treatment method (radical prostatectomy or radiotherapy). DNA will be extracted from archived tissue (formalin-fixed paraffin embedded - FFPE) for all biological specimens - either in dominant lesion in radical prostatectomy or diagnostic prostate biopsy and metastasis, using approved protocol for nucleic acid extraction. Availability of radical prostatectomy specimen and largest metastasis would allow for significant amounts of tissue for initial whole exome sequencing (WES) of the primary tumor and metastasis (200x deep sequencing relative to 30x normal blood DNA sequencing). The plan is to obtain tissue from the same metastasis after onset of castrate resistance (if clinically available) as well. Bioinformatics analyses will be performed to obtain panel of genomic changes encompassing whole disease spectrum. The investigators will then compare all these clonal signals to determine if these metastatic clones were present in primary tumor at the time of the initial diagnosis, prior to any treatment and if treatment-resistant clones were present early, before initiation of therapy for metastatic disease. This will test the concept of treatment (ADT)-induced selection versus adaptation during a course of ADT and develop novel signatures of SNV, CNV and GRs within two levels of metastases that have not yet been clearly defined.

(ii) Aim 4, 5: Comparative analysis between DNA profile of primary tumor and metastases, so this project might augment knowledge on site-specific signature(s) predictive for this outcome in highly heterogeneous population of prostate cancer patients.

Translational relevance

The results generated from the proposed work might be relevant in the push towards personalised therapies in prostate cancer patient's management. Currently, there is no personalized approach in this area as all patients are being treated in the same manner regardless of underlying biology of the disease. In the case example of metastatic prostate cancer where ADT is primary treatment modality, there is a potential for clinical utility of genomic signature that predicts failure to hormonal therapy and gives insight of driving mutations of disease progression, from primary tumor to metastases. Finally, relevant data will be gathered on feasibility of genomic testing in the multimodal management of patients with metastatic prostate cancer for the first time in Croatia. There is also a point of assessing utility of obtained genetic information for presumable use of targeted therapies and making treatment decisions in the real-world clinical setting in transitional eastern European country with emerging pharmaceutical market.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with newly diagnosed metastatic prostate cancer
2. Androgen dependent disease measured by declining PSA
3. ECOG PS 0 or 1
4. Life-expectancy based on comorbid conditions >2 years
5. Ability to understand and willingness to sign informed consent
6. Must be candidate for radiation therapy

Exclusion Criteria:

1. Poor performance status, history of connective tissue disorder
2. Psychiatric or medical conditions which would not allow the patient to undergo the proposed treatment safely
3. Known brain metastasis

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival | 4 years
  Time to prostate specific antigen (PSA) progression

SECONDARY OUTCOMES:
Prostate, bone marrow and viscera progression-free survival | 4 years
  Number of participants with radiographic disease progression in prostate, bone and visceral organs
Expression of integrins | 4 years
  Number of participants with expression of analysed genes : 2 housekeeping genes; integrin subunits αv, β3, β5, α4β1 ; 3 EMT markers N-cadherin, E-cadherin, vimentin before radiotherapy, after radiotherapy and at the time of the disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fröbe, MD, PhD, Principal Investigator — UHC Sestre Milosrdnice, Department of Oncology and Nuclear Medicine, Vinogradska 29, 10 000 Zagreb, Croatia
Locations (1):
- Ana Frobe, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Culp SH, Schellhammer PF, Williams MB. Might men diagnosed with metastatic prostate cancer benefit from definitive treatment of the primary tumor? A SEER-based study. Eur Urol. 2014 Jun;65(6):1058-66. doi: 10.1016/j.eururo.2013.11.012. Epub 2013 Nov 20. PMID 24290503
- [Result] Fossati N, Trinh QD, Sammon J, Sood A, Larcher A, Sun M, Karakiewicz P, Guazzoni G, Montorsi F, Briganti A, Menon M, Abdollah F. Identifying optimal candidates for local treatment of the primary tumor among patients diagnosed with metastatic prostate cancer: a SEER-based study. Eur Urol. 2015 Jan;67(1):3-6. doi: 10.1016/j.eururo.2014.08.056. Epub 2014 Sep 10. PMID 25217422
- [Result] Gratzke C, Engel J, Stief CG. Role of radical prostatectomy in metastatic prostate cancer: data from the Munich Cancer Registry. Eur Urol. 2014 Sep;66(3):602-3. doi: 10.1016/j.eururo.2014.04.009. Epub 2014 May 10. No abstract available. PMID 24821581
- [Result] Psaila B, Lyden D. The metastatic niche: adapting the foreign soil. Nat Rev Cancer. 2009 Apr;9(4):285-93. doi: 10.1038/nrc2621. PMID 19308068
- [Result] Ganguly SS, Li X, Miranti CK. The host microenvironment influences prostate cancer invasion, systemic spread, bone colonization, and osteoblastic metastasis. Front Oncol. 2014 Dec 15;4:364. doi: 10.3389/fonc.2014.00364. eCollection 2014. PMID 25566502
- [Result] Shinka T, Onodera D, Tanaka T, Shoji N, Miyazaki T, Moriuchi T, Fukumoto T. Serotonin synthesis and metabolism-related molecules in a human prostate cancer cell line. Oncol Lett. 2011 Mar;2(2):211-215. doi: 10.3892/ol.2011.244. Epub 2011 Jan 20. PMID 22866066
- [Result] Dizeyi N, Bjartell A, Nilsson E, Hansson J, Gadaleanu V, Cross N, Abrahamsson PA. Expression of serotonin receptors and role of serotonin in human prostate cancer tissue and cell lines. Prostate. 2004 May 15;59(3):328-36. doi: 10.1002/pros.10374. PMID 15042609
- [Result] Widmark A, Klepp O, Solberg A, Damber JE, Angelsen A, Fransson P, Lund JA, Tasdemir I, Hoyer M, Wiklund F, Fossa SD; Scandinavian Prostate Cancer Group Study 7; Swedish Association for Urological Oncology 3. Endocrine treatment, with or without radiotherapy, in locally advanced prostate cancer (SPCG-7/SFUO-3): an open randomised phase III trial. Lancet. 2009 Jan 24;373(9660):301-8. doi: 10.1016/S0140-6736(08)61815-2. Epub 2008 Dec 16. PMID 19091394
- [Result] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- See also: Integrins in Prostate Cancer Invasion and Metastasis — http://dx.doi.org/10.5772/53482